CLINICAL TRIAL: NCT02576288
Title: Effects of Sitagliptin on Arterial Vasoreactivity and Proatherogenic Mediators in Obesity
Brief Title: Sitagliptin Effects on Arterial Vasculature and Inflammation in Obesity
Acronym: SAVORO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Fred Sattler, MD, Professor of Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-13-00345
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Atherosclerosis; Inflammation
Keywords: Sitagliptin; Brachial artery flow mediated dilation; Carotid stiffness; Pro-inflammatory; Pro-atherogenic; M1 macrophages
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental): 100mg will be administered by mouth daily for 28days
  Interventions: Drug: Sitagliptin
- Matching Placebo (Placebo Comparator): One placebo will be administered by mouth daily for 28days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — anti-inflammatory properties
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — No anti-inflammatory properties
  Other Names: Dummy pill
  Arms: Matching Placebo

SUMMARY:
Abdominal obesity is a major risk factor for heart attack, stroke, peripheral vascular disease, dementia, cancer and Type 2 diabetes. The central hypothesis for this proposal is that pro-atherogenic mediators emanate from inflammation in deep subcutaneous adipose tissue (dSAT) that are released into the systemic circulation and damage the arterial vasculature. The investigators postulate that inflammation of dSAT, when quantified by macrophage phenotyping/enumeration will be a) closely linked with systemic levels of pro-atherogenic mediators and b) tightly associated with endothelial dysfunction and loss of central arterial elasticity, which are highly predictive of future cardiovascular disease (CVD) complications. These relationships provide the basis for macrophage-targeted therapy to reduce obesity-related inflammation and impaired arterial vasoreactivity. The investigators will evaluate a novel approach using a dipeptidyl peptidase 4 inhibitor (DPP4i) sitagliptin, which blocks signal transduction for monocyte/macrophage activation. Thus, in abdominally obese, 18-40 years-old adults without clinical CVD, the show study is expected to show that sitagliptin versus placebo will:

1. significantly improve early measures of arterial damage (brachial artery endothelial dysfunction and reduced carotid elasticity).
2. significantly attenuate inflammation in dSAT and local production of pro-inflammatory mediators in adipose tissue, which will be associated with decreases in systemic pro-atherogenic mediators that contribute to atherogenesis.

Since many obese persons fail to sustain weight loss by lifestyle interventions including diet and exercise, an important public health goal is to identify relatively safe alternative strategies that can be used pre-emptively in "asymptomatic" obese persons when arterial dysfunction and damage is still reversible before atherosclerosis progresses to serious CVD events.

DETAILED DESCRIPTION:
APPROACH:

Overview of Study Design: This is a double-masked, randomized, placebo-controlled pilot study of treatment sitagliptin (100mg/day) to suppress monocyte/macrophage activation in obese non-diabetic participants. 16 abdominally obese18-40 year-old largely minorities will be randomized 3:1 to receive sitagliptin (N=12) or matching placebo (N=4) daily for 28 days.

Eligibility Criteria for the Study Cohort: Based on prior studies conducted by the investigators, approximately 60-70% of participants enrolled will be Hispanics and African Americans. Both minorities have increased prevalence of insulin resistance (IR) at young ages. In their prior studies, insulin resistance (HOMA-IR* ≥3.0) had a predictive value of 88% for crown like structure in abdominal fat (a surrogate for fat inflammation); the inclusion criterion for IR will assure that most study subjects will have abdominal fat inflammation.

* homeostatic method of analysis-insulin resistance

Inclusion Criteria

1. Age 18-40 years of age
2. Stable weight (no change >3% in prior 6 months)
3. Waist circumference ≥102cm for men; ≥88cm for women
4. Fasting plasma glucose 100-125, HgbA1C 5.7-6.4% or HOMA-IR* ≥3.0

Exclusion Criteria:

1. Regular use of a non-steroidal anti-inflammatory drug (NSAID); unwilling to stop NSAID drug
2. On statin or other prescription anti-inflammatory drugs
3. Diabetes or clinically evident cardiovascular disease
4. Smoking daily or consuming >200g alcohol/day

Study participants will be adults 18-40 years of age to exclude older persons with irreversible atherosclerosis (e.g. calcified, stenotic plaque) or subclinical arterial thrombus which release inflammatory mediators. Persons with Type 2 diabetes (a myocardial infarction equivalent) and those receiving "statins" (also potent anti-inflammatory drugs) will be excluded, thereby further excluding participants with advanced atherosclerosis. The goal is to identify and study persons with abdominal obesity and inflammation at a younger age as a potential target population for pre-emptive anti-inflammatory therapy to prevent serious CVD events over ensuing years.

Outcome Measures:

1. Change in arterial vasoreactivity measured and quantified by ultrasound assessment of brachial artery flow mediated dilation and carotid stiffness (elasticity and distensibility).
2. Change in measures of inflammation in intra-abdominal adipose tissue:

   1. M1 pro-inflammatory macrophages and M2 anti-inflammatory macrophages by fluorescent activated cell sorting.
   2. Ex vivo secretion of inflammatory mediators from macrophages fractions.
3. Change in systemic pro-inflammatory/pro-atherogenic markers and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* abdominal obesity (≥102cm for men and ≥88cm for women)
* impaired glucose tolerance with fasting plasma glucose 100-125 or HgbA1C 5.7-6.4%
* insulin resistance with HOMA-IR ≥3.0
* stable weight with no change >3% in prior 6 months

Exclusion Criteria:

* regular use of non-steroidal anti-inflammatory drug and unwilling to stop
* on statin or other anti-inflammatory medication or herbal remedy
* diabetes or clinically evident cardiovascular disease
* smoking daily or consuming >200g of alcohol daily
* active renal, hepatic, rheumatological or infectious disorder within 28 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Ultrasound quantification of change in brachial artery flow mediated dilation and carotid stiffness (elasticity and distensibility) | Immediately before and after 28 days of study thearpy
  To ascertain effects of sitagliptin vs placebo on endothelial function (brachial artery flow) and structural measure of atherosclerosis (carotid stiffness)

SECONDARY OUTCOMES:
Deep subcutaneous adipose tissue inflammation | Immediately before and after 28 days of study thearpy
  quantify M1 and M2 macrophages by fluorescence activated cell sorting and ex vivo secretion of pro-inflammatory mediators

OTHER OUTCOMES:
Systemic markers of inflammation/atherogenic mediators and insulin resistance | Immediately before and after 28 days of study thearpy
  To ascertain if sitagliptin vs placebo will decrease C-reactive protein, Tumor Necrosis Factor alpha, interleukin 6, soluble CD40 ligand, interferon like protein 10, IP-10, homeostatic method of assessment for insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Sattler, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California Health Sciences Campus, Los Angeles, California, United States